CLINICAL TRIAL: NCT01984242
Title: A Phase II, Randomized Study of Atezolizumab (Anti-PD-L1 Antibody) Administered as Monotherapy or in Combination With Bevacizumab Versus Sunitinib in Patients With Untreated Advanced Renal Cell Carcinoma
Brief Title: A Study of Atezolizumab (an Engineered Anti-Programmed Death-Ligand 1 [PD-L1] Antibody) as Monotherapy or in Combination With Bevacizumab (Avastin®) Compared to Sunitinib (Sutent®) in Participants With Untreated Advanced Renal Cell Carcinoma
Acronym: IMmotion150
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO29074; 2013-003167-58 (EudraCT Number)
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Results first posted 2017-12-21 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — atezolizumab; Bevacizumab; Sunitinib

ARMS (3):
- Atezolizumab and Bevacizumab (Experimental): Atezolizumab 1200 milligrams (mg) and bevacizumab 15 milligrams per kilogram (mg/kg) will be administered as intravenous (IV) infusions every 3 weeks (q3w) on Day 1 and Day 22 of each 6-week cycle until disease progression.
  Interventions: Drug: Atezolizumab (MPDL3280A), an Engineered Anti-PD-L1 Antibody; Drug: Bevacizumab
- Atezolizumab (Experimental): Atezolizumab 1200 mg will be administered as IV infusion q3w on Day 1 and Day 22 of each 6-week cycle until disease progression. Upon disease progression, participants (except European Union [EU] participants) can crossover to receive atezolizumab and bevacizumab combination until disease progression, lack of clinical benefit, unacceptable toxicity, withdrawal from study, or study completion or termination.
  Interventions: Drug: Atezolizumab (MPDL3280A), an Engineered Anti-PD-L1 Antibody; Drug: Bevacizumab
- Sunitinib (Active Comparator): Sunitinib 50 mg will be administered orally once daily on Days 1 to 28 of each 6-week cycle until disease progression. Upon disease progression, participants can crossover to receive atezolizumab and bevacizumab combination until disease progression, lack of clinical benefit, unacceptable toxicity, withdrawal from study, or study completion or termination.
  Interventions: Drug: Atezolizumab (MPDL3280A), an Engineered Anti-PD-L1 Antibody; Drug: Bevacizumab; Drug: Sunitinib

INTERVENTIONS:
Drug: Atezolizumab (MPDL3280A), an Engineered Anti-PD-L1 Antibody — Atezolizumab will be administered according to the dosage schedule mentioned in the arm description.
  Other Names: Tecentriq; MPDL3280A; RO5541267
Drug: Bevacizumab — Bevacizumab will be administered according to the dosage schedule mentioned in the arm description.
  Other Names: Avastin
Drug: Sunitinib — Sunitinib will be administered according to the dosage schedule mentioned in the arm description.
  Other Names: Sutent
  Arms: Sunitinib

SUMMARY:
This multicenter, randomized, open-label study will evaluate the efficacy, safety and tolerability of atezolizumab as monotherapy or in combination with bevacizumab versus sunitinib in participants with histologically confirmed, inoperable, locally advanced or metastatic renal cell carcinoma who have not received prior systemic therapy either in the adjuvant or metastatic setting.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable advanced or metastatic renal cell carcinoma with component of clear cell histology and/or component of sarcomatoid histology that has not been previously treated with any systemic agents, including treatment in the adjuvant setting
* Measurable disease, as defined by RECIST v1.1
* Karnofsky performance score greater than or equal to (>/=) 70
* Adequate hematologic and end-organ function as defined by protocol
* Women of childbearing potential and male participants with partners of childbearing potential must agree to use highly effective methods of contraception as defined by protocol

Exclusion Criteria:

Disease-Specific Exclusions:

* Radiotherapy for renal cell carcinoma within 14 days prior to Cycle 1, Day 1 with the exception of single-fraction radiotherapy given for the indication of pain control
* Known active malignancies or metastasis of the brain or spinal cord or leptomeningeal disease, as determined by computed tomography (CT) or magnetic resonance imaging (MRI) evaluation during screening and prior radiographic assessments
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)
* Uncontrolled hypercalcemia or symptomatic hypercalcemia
* Malignancies other than renal cell carcinoma within 5 years prior to Cycle 1, Day 1, with the exception of those with a negligible risk of metastasis or death, treated with expected curative outcome

General Medical Exclusions:

* Life expectancy of less than (<) 12 weeks
* Pregnant and lactating women
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* History of autoimmune disease
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
* Participants with active or chronic hepatitis B, active hepatitis C, Human Immunodeficiency Virus (HIV) positive test, significant cardiovascular disease
* Prior allogeneic stem cell or solid organ transplant

Exclusion Criteria Related to Medications:

* Prior treatment with Cluster of Differentiation 137 (CD137) agonists, anti-Cytotoxic T-Lymphocyte Antigen-4 (anti-CTLA-4), anti-programmed death-1 (anti-PD-1), or anti-PD-L1 therapeutic antibody or pathway-targeting agents
* Treatment with systemic immunostimulatory agents for any reason within 6 weeks or five half-lives of the drug, whichever is shorter, prior to Cycle 1, Day 1
* Treatment with systemic immunosuppressive medications within 2 weeks prior to Cycle 1, Day 1

Bevacizumab- and Sunitinib-Specific Exclusions:

* Inadequately controlled hypertension
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association Class II or greater congestive heart failure
* History of myocardial infarction or unstable angina, stroke or transient ischemic attack within 3 months prior to Cycle 1, Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2014-01-08 (Actual); Primary Completion 2016-10-17 (Actual); Study Completion 2019-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (45):
- United States (25):
  - HonorHealth Research Institute - Bisgrove, Scottsdale, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCLA, Los Angeles, California
  - University of California, San Francisco, California
  - Univ Colorado Health Sci Ctr, Aurora, Colorado
  - Rocky Mountain Cancer Ctr - Denver (Williams), Denver, Colorado
  - Yale Uni School of Medicine; Section of Medical Oncology, New Haven, Connecticut
  - Georgetown U; Lombardi Comp Can, Washington D.C., District of Columbia
  - SCRI Florida Cancer Specialists South, Fort Myers, Florida
  - Mayo Clinic-Jacksonville, Jacksonville, Florida
  - Florida Cancer Specialist, North Region, St. Petersburg, Florida
  - The University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Inst., Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Karmanos Cancer Institute., Detroit, Michigan
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Memorial Sloan-Kettering, New York, New York
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Cleveland Clinic Foundation; Taussig Cancer Center, Cleveland, Ohio
  - Oncology Associates of Oregon, P.C, Eugene, Oregon
  - Northwest Cancer Specialists, P.C., Tigard, Oregon
  - Tennessee Oncology PLLC - Nashville (20th Ave), Nashville, Tennessee
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Texas Oncology-Baylor Sammons Cancer Center, Dallas, Texas
- Fakultni nemocnice Olomouc, Olomouc, Czechia
- France (3):
  - Hopital Europeen Georges Pompidou; Service D'Oncologie Medicale, Paris
  - CHU Bordeaux, Pessac
  - Institut Gustave Roussy; Departement Oncologie Medicale, Villejuif
- Germany (3):
  - Medizinische Hochschule; Zentrum Innere Medizin; Abt. Hämatologie u. Onkologie, Hanover
  - Klinikum d.Universität München Campus Großhadern, München
  - Klinikum rechts der Isar der TU München; Klinikapotheke, München
- Italy (3):
  - Irccs Istituto Nazionale Dei Tumori (Int);S.C. Medicina Oncologica 2, Milan, Lombardy
  - Medical Oncology, Arezzo, Arezzo, Tuscany
  - Azienda Ospedaliera Universitaria Senese, U.O.C. Immunoterapia Oncologica, Siena, Tuscany
- Centrum Med. Ostrobramska NZOZ Magodent, Warsaw, Poland
- Romania (2):
  - Prof. Dr. I. Chiricuta Institute of Oncology, Cluj-Napoca
  - Medisprof SRL, Cluj-Napoca
- Spain (4):
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona. Unidad de Nuevas Terapias;Oncology Department, Barcelona
  - Hosp de Madrid Norte Sanchinarro; Centro Integral; Onco Clara Campal, Madrid
- United Kingdom (3):
  - Barts and the London NHS Trust., London
  - Royal Marsden Hospital - London, London
  - Christie Hospital Nhs Trust; Medical Oncology, Manchester

REFERENCES:
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] Pal SK, McDermott DF, Atkins MB, Escudier B, Rini BI, Motzer RJ, Fong L, Joseph RW, Oudard S, Ravaud A, Bracarda S, Suarez C, Lam ET, Choueiri TK, Ding B, Quach C, Hashimoto K, Schiff C, Piault-Louis E, Powles T. Patient-reported outcomes in a phase 2 study comparing atezolizumab alone or with bevacizumab vs sunitinib in previously untreated metastatic renal cell carcinoma. BJU Int. 2020 Jul;126(1):73-82. doi: 10.1111/bju.15058. Epub 2020 Apr 24. PMID 32233107

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 305 participants enrolled in this study. Participants enrolled in atezolizumab (except European Union [EU] participants) or sunitinib group could crossover to receive atezolizumab and bevacizumab combination therapy in case of disease progression. Some participants didn't complete due to study termination, but study was completed as planned.
Groups:
- Atezolizumab and Bevacizumab: Atezolizumab 1200 milligrams (mg) and bevacizumab 15 milligrams per kilogram (mg/kg) were administered as intravenous (IV) infusions every 3 weeks (q3w) on Day 1 and Day 22 of each 6-week cycle until disease progression.
- Atezolizumab: Atezolizumab 1200 mg was administered as IV infusion q3w on Day 1 and Day 22 of each 6-week cycle until disease progression. Upon disease progression, participants (except EU participants) could crossover to receive atezolizumab and bevacizumab combination until disease progression, lack of clinical benefit, unacceptable toxicity, withdrawal from study, or study completion or termination.
- Sunitinib: Sunitinib 50 mg was administered orally once daily on Days 1 to 28 of each 6-week cycle until disease progression. Upon disease progression, participants could crossover to receive atezolizumab and bevacizumab combination until disease progression, lack of clinical benefit, unacceptable toxicity, withdrawal from study, or study completion or termination.
Period: Overall Study
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Started | 101 | 103 | 101
Treated | 101 | 103 | 100
Completed | 0 | 0 | 0
Not Completed | 101 | 103 | 101
Not completed — Death | 52 | 50 | 52
Not completed — Withdrawal by Subject | 5 | 3 | 10
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Lost to Follow-up | 4 | 0 | 3
Not completed — Sponsor Decision | 1 | 0 | 0
Not completed — Non-Compliance | 1 | 0 | 0
Not completed — Study terminated by Sponsor | 38 | 50 | 34
Not completed — Disease Progression | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants regardless of whether they received any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib | Total
Number analyzed (Participants) | 101 | 103 | 101 | 305
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (10.8) | 60.1 (10.2) | 59.7 (10.8) | 60.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 26 | 22 | 75
  Male | 74 | 77 | 79 | 230

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease Progression Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) Via Independent Review Committee (IRC) Assessment or Death in Intent-to-Treat (ITT) Population
Description: Progressive Disease (PD): at least a 20 percent (%) increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline, and an absolute increase of at least 5 millimeters (mm); appearance of one or more new target or non-target lesions; or unequivocal progression of existing non-target lesions.
Time Frame: From randomization until disease progression or death due to any cause (until data cut-off date 17 October 2016, up to approximately 2.75 years)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 101 | 103 | 101
percentage of participants | 66.3 | 59.2 | 58.4

2. Primary Outcome: Progression-Free Survival (PFS) Per RECIST v1.1 Via IRC Assessment in ITT Population
Description: PFS was defined as the time from randomization to the first occurrence of PD or death due to any cause. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline, and an absolute increase of at least 5 mm; appearance of one or more new target or non-target lesions; or unequivocal progression of existing non-target lesions. Kaplan-Meier methodology was used to estimate PFS.
Time Frame: as for outcome 1
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 101 | 103 | 101
months | 11.7 [8.4 to 17.3] | 6.1 [5.4 to 13.6] | 8.4 [7.0 to 14.0]
Statistical Analysis 1: Comparison: Atezolizumab and Bevacizumab vs Sunitinib; Test type: Superiority; p = 0.9819, Log Rank; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.69 to 1.45]
Statistical Analysis 2: Comparison: Atezolizumab vs Sunitinib; Test type: Superiority; p = 0.3580, Log Rank; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.82 to 1.71]

3. Primary Outcome: Percentage of Participants With Disease Progression Per RECIST v1.1 Via IRC Assessment or Death in Immune Cell 1/2/3 (IC1/2/3) Population
Description: PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline, and an absolute increase of at least 5 mm; appearance of one or more new target or non-target lesions; or unequivocal progression of existing non-target lesions.
Time Frame: as for outcome 1
Population: IC1/2/3 population included ITT participants with programmed death-ligand 1 (PD-L1) expression of greater than or equal to (>=) 1% on tumor-infiltrating immune cells.
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 50 | 54 | 60
percentage of participants | 58.0 | 59.3 | 68.3

4. Primary Outcome: PFS Per RECIST v1.1 Via IRC Assessment in IC1/2/3 Population
Description: as for outcome 2
Time Frame: as for outcome 1
Population: IC1/2/3 population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 50 | 54 | 60
months | 14.7 [8.2 to 25.1] | 5.5 [3.0 to 13.9] | 7.8 [3.8 to 10.8]
Statistical Analysis 1: Comparison: Atezolizumab and Bevacizumab vs Sunitinib; Test type: Superiority; p = 0.0952, Log Rank; Hazard Ratio (HR) = 0.64, 95% CI [0.38 to 1.08]
Statistical Analysis 2: Comparison: Atezolizumab vs Sunitinib; Test type: Superiority; p = 0.9172, Log Rank; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.63 to 1.67]

5. Secondary Outcome: Percentage of Participants With Disease Progression Per RECIST v1.1 Via IRC Assessment or Death in Participants Who Have Tumors With Higher Than Median Expression of an Immune Gene Signature
Description: as for outcome 3
Time Frame: as for outcome 1
Population: Biomarker evaluable population included ITT participants whose tumor samples had sufficient material available for gene signature expression analyses. Participants with higher than median expression of an immune gene signature were included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 45 | 44 | 42
percentage of participants | 55.6 | 61.4 | 73.8

6. Secondary Outcome: PFS Per RECIST v1.1 Via IRC Assessment in Participants Who Have Tumors With Higher Than Median Expression of an Immune Gene Signature
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Biomarker evaluable population. Participants with higher than median expression of an immune gene signature were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 45 | 44 | 42
months | 17.5 [10.3 to NA] — Data could not be estimated due to high number of censored participants. | 5.7 [3.2 to 16.7] | 7.1 [4.2 to 8.7]
Statistical Analysis 1: Comparison: Atezolizumab and Bevacizumab vs Sunitinib; Test type: Superiority; p = 0.0153, Log Rank; Hazard Ratio (HR) = 0.48, 95% CI 2-sided [0.26 to 0.87]
Statistical Analysis 2: Comparison: Atezolizumab vs Sunitinib; Test type: Superiority; p = 0.5545, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.48 to 1.46]

7. Secondary Outcome: Percentage of Participants With Disease Progression Per RECIST v1.1 Via Investigator Assessment or Death in Participants Who Have Tumors With Higher Than Median Expression of an Immune Gene Signature
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 45 | 44 | 42
percentage of participants | 57.8 | 77.3 | 83.3

8. Secondary Outcome: PFS Per RECIST v1.1 Via Investigator Assessment in Participants Who Have Tumors With Higher Than Median Expression of an Immune Gene Signature
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 45 | 44 | 42
months | 16.6 [8.2 to NA] — Data could not be estimated due to high number of censored participants. | 5.5 [3.0 to 11.1] | 6.8 [5.4 to 8.7]
Statistical Analysis 1: Comparison: Atezolizumab and Bevacizumab vs Sunitinib; Test type: Superiority; p = 0.0086, Log Rank; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.28 to 0.84]
Statistical Analysis 2: Comparison: Atezolizumab vs Sunitinib; Test type: Superiority; p = 0.7675, Log Rank; Hazard Ratio (HR) = 0.93, 95% CI [0.56 to 1.53]

9. Secondary Outcome: Percentage of Participants With Disease Progression Per RECIST v1.1 Via IRC Assessment or Death in Participants Who Have Tumors With Higher Than the 33rd Percentile Expression of an Immune Gene Signature
Description: as for outcome 3
Time Frame: as for outcome 1
Population: Biomarker evaluable population. Participants with higher than the 33rd percentile expression of an immune gene signature were included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 61 | 55 | 60
percentage of participants | 59.0 | 58.2 | 65.0

10. Secondary Outcome: PFS Per RECIST v1.1 Via IRC Assessment in Participants Who Have Tumors With Higher Than the 33rd Percentile Expression of an Immune Gene Signature
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 61 | 55 | 60
months | 13.8 [8.3 to 25.1] | 5.7 [5.4 to 17.3] | 8.2 [5.7 to 11.4]
Statistical Analysis 1: Comparison: Atezolizumab and Bevacizumab vs Sunitinib; Test type: Superiority; p = 0.1973, Log Rank; Hazard Ratio (HR) = 0.72, 95% CI [0.44 to 1.18]
Statistical Analysis 2: Comparison: Atezolizumab vs Sunitinib; Test type: Superiority; p = 0.7738, Log Rank; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.65 to 1.76]

11. Secondary Outcome: Percentage of Participants With Disease Progression Per RECIST v1.1 Via Investigator Assessment or Death in Participants Who Have Tumors With Higher Than the 33rd Percentile Expression of an Immune Gene Signature
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 61 | 55 | 60
percentage of participants | 63.9 | 76.4 | 78.3

12. Secondary Outcome: PFS Per RECIST v1.1 Via Investigator Assessment in Participants Who Have Tumors With Higher Than the 33rd Percentile Expression of an Immune Gene Signature
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 61 | 55 | 60
months | 11.1 [8.1 to 19.3] | 5.5 [3.0 to 10.9] | 7.1 [5.8 to 11.3]
Statistical Analysis 1: Comparison: Atezolizumab and Bevacizumab vs Sunitinib; Test type: Superiority; p = 0.0830, Log Rank; Hazard Ratio (HR) = 0.68, 95% CI [0.43 to 1.06]
Statistical Analysis 2: Comparison: Atezolizumab vs Sunitinib; Test type: Superiority; p = 0.7141, Log Rank; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.70 to 1.69]

13. Secondary Outcome: Percentage of Participants With Disease Progression Per RECIST v1.1 Via Investigator Assessment or Death in ITT Population
Description: as for outcome 3
Time Frame: as for outcome 1
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 101 | 103 | 101
percentage of participants | 71.3 | 75.7 | 75.2

14. Secondary Outcome: PFS Per RECIST v1.1 Via Investigator Assessment in ITT Population
Description: as for outcome 2
Time Frame: as for outcome 1
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 101 | 103 | 101
months | 11.1 [8.2 to 13.5] | 5.5 [3.0 to 8.4] | 7.8 [5.7 to 11.2]
Statistical Analysis 1: Comparison: Atezolizumab and Bevacizumab vs Sunitinib; Test type: Superiority; p = 0.2541, Log Rank; Hazard Ratio (HR) = 0.82, 95% CI [0.59 to 1.15]
Statistical Analysis 2: Comparison: Atezolizumab vs Sunitinib; Test type: Superiority; p = 0.3103, Log Rank; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.86 to 1.63]

15. Secondary Outcome: Percentage of Participants With Disease Progression Per RECIST v1.1 Via Investigator Assessment or Death in IC1/2/3 Population
Description: as for outcome 3
Time Frame: as for outcome 1
Population: IC1/2/3 population
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 50 | 54 | 60
percentage of participants | 66.0 | 74.1 | 81.7

16. Secondary Outcome: PFS Per RECIST v1.1 Via Investigator Assessment in IC1/2/3 Population
Description: as for outcome 2
Time Frame: as for outcome 1
Population: IC1/2/3 population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 50 | 54 | 60
months | 11.1 [8.1 to 16.7] | 5.5 [3.0 to 10.9] | 7.0 [5.6 to 11.2]
Statistical Analysis 1: Comparison: Atezolizumab and Bevacizumab vs Sunitinib; Test type: Superiority; p = 0.0351, Log Rank; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.37 to 0.97]
Statistical Analysis 2: Comparison: Atezolizumab vs Sunitinib; Test type: Superiority; p = 0.9769, Log Rank; Hazard Ratio (HR) = 0.99, 95% CI [0.64 to 1.54]

17. Secondary Outcome: Percentage of Participants With Objective Response (Complete Response [CR] or Partial Response [PR]) Per RECIST v1.1 Via IRC Assessment in ITT Population
Description: Objective Response was defined as CR or PR. CR: disappearance of all target and non-target lesions and (if applicable) normalization of tumor marker level; or reduction in short axis of any pathological lymph nodes (whether target or non-target) to less than (<) 10 mm. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters; or persistence of one or more non-target lesion(s) and/or (if applicable) maintenance of tumor marker level above the normal limits.
Time Frame: as for outcome 1
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 101 | 103 | 101
percentage of participants | 31.7 [22.78 to 41.69] | 25.2 [17.20 to 34.76] | 28.7 [20.15 to 38.57]
Statistical Analysis 1: Comparison: Atezolizumab and Bevacizumab vs Sunitinib; Test type: Superiority; p = 0.6492, Cochran-Mantel-Haenszel; Difference in response rates = 2.97, 95% CI 2-sided [-10.68 to 16.62]
Statistical Analysis 2: Comparison: Atezolizumab vs Sunitinib; Test type: Superiority; p = 0.5433, Cochran-Mantel-Haenszel; Difference in response rates = -3.47, 95% CI [-16.63 to 9.69]

18. Secondary Outcome: Percentage of Participants With Objective Response Per RECIST v1.1 Via IRC Assessment in IC1/2/3 Population
Description: Objective Response was defined as CR or PR. CR: disappearance of all target and non-target lesions and (if applicable) normalization of tumor marker level; or reduction in short axis of any pathological lymph nodes (whether target or non-target) to <10 mm. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters; or persistence of one or more non-target lesion(s) and/or (if applicable) maintenance of tumor marker level above the normal limits.
Time Frame: as for outcome 1
Population: IC1/2/3 population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 50 | 54 | 60
percentage of participants | 46.0 [31.81 to 60.68] | 27.8 [16.46 to 41.64] | 26.7 [16.07 to 39.66]
Statistical Analysis 1: Comparison: Atezolizumab and Bevacizumab vs Sunitinib; Test type: Superiority; p = 0.0141, Cochran-Mantel-Haenszel; Difference in response rates = 19.33, 95% CI 2-sided [-0.28 to 38.94]
Statistical Analysis 2: Comparison: Atezolizumab vs Sunitinib; Test type: Superiority; p = 0.8719, Cochran-Mantel-Haenszel; Difference in response rates = 1.11, 95% CI 2-sided [-17.02 to 19.24]

19. Secondary Outcome: Percentage of Participants With Objective Response Per RECIST v1.1 Via Investigator Assessment in ITT Population
Description: as for outcome 18
Time Frame: as for outcome 1
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 101 | 103 | 101
percentage of participants | 34.7 [25.46 to 44.77] | 23.3 [15.54 to 32.66] | 32.7 [23.67 to 42.72]
Statistical Analysis 1: Comparison: Atezolizumab and Bevacizumab vs Sunitinib; Test type: Superiority; p = 0.8068, Cochran-Mantel-Haenszel; Difference in response rates = 1.98, 95% CI 2-sided [-12.04 to 16.00]
Statistical Analysis 2: Comparison: Atezolizumab vs Sunitinib; Test type: Superiority; p = 0.1321, Cochran-Mantel-Haenszel; Difference in response rates = -9.37, 95% CI [-22.61 to 3.87]

20. Secondary Outcome: Percentage of Participants With Objective Response Per RECIST v1.1 Via Investigator Assessment in IC1/2/3 Population
Description: as for outcome 18
Time Frame: as for outcome 1
Population: IC1/2/3 population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 50 | 54 | 60
percentage of participants | 48.0 [33.66 to 62.58] | 25.9 [14.96 to 39.65] | 28.3 [17.45 to 41.44]
Statistical Analysis 1: Comparison: Atezolizumab and Bevacizumab vs Sunitinib; Test type: Superiority; p = 0.0199, Cochran-Mantel-Haenszel; Difference in response rates = 19.67, 95% CI 2-sided [-0.10 to 39.44]
Statistical Analysis 2: Comparison: Atezolizumab vs Sunitinib; Test type: Superiority; p = 0.7836, Cochran-Mantel-Haenszel; Difference in response rates = -2.41, 95% CI 2-sided [-20.50 to 15.68]

21. Secondary Outcome: Percentage of Participants With Objective Response Per Modified RECIST Via Investigator Assessment in ITT Population
Description: Objective Response was defined as CR or PR. CR: disappearance of all target and non-target lesions; or reduction in short axis of any pathological lymph nodes (whether target or non-target) to <10 mm. PR: at least a 30% decrease in the sum of diameters of target and all new measurable lesions, taking as reference the baseline sum of diameters, in absence of CR.
Time Frame: as for outcome 1
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 101 | 103 | 101
percentage of participants | 37.6 [28.18 to 47.82] | 25.2 [17.20 to 34.76] | 33.7 [24.56 to 43.75]
Statistical Analysis 1: Comparison: Atezolizumab and Bevacizumab vs Sunitinib; Test type: Superiority; p = 0.6231, Cochran-Mantel-Haenszel; Difference in response rates = 3.96, 95% CI 2-sided [-10.23 to 18.15]
Statistical Analysis 2: Comparison: Atezolizumab vs Sunitinib; Test type: Superiority; p = 0.1816, Cochran-Mantel-Haenszel; Difference in response rates = -8.42, 95% CI 2-sided [-21.86 to 5.02]

22. Secondary Outcome: Percentage of Participants With Objective Response Per Modified RECIST Via Investigator Assessment in IC1/2/3 Population
Description: as for outcome 21
Time Frame: as for outcome 1
Population: IC1/2/3 population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 50 | 54 | 60
percentage of participants | 52.0 [37.42 to 66.34] | 27.8 [16.46 to 41.64] | 30.0 [18.85 to 43.21]
Statistical Analysis 1: Comparison: Atezolizumab and Bevacizumab vs Sunitinib; Test type: Superiority; p = 0.0111, Cochran-Mantel-Haenszel; Difference in response rates = 22.00, 95% CI 2-sided [2.11 to 41.89]
Statistical Analysis 2: Comparison: Atezolizumab vs Sunitinib; Test type: Superiority; p = 0.8209, Cochran-Mantel-Haenszel; Difference in response rates = -2.22, 95% CI 2-sided [-20.63 to 16.19]

23. Secondary Outcome: Percentage of Participants With Disease Progression Per Modified RECIST Via Investigator Assessment or Death in ITT Population
Description: PD: at least a 20% increase in the sum of diameters of all target and new measurable lesions, taking as reference the smallest sum on study, including baseline, and an absolute increase of at least 5 mm.
Time Frame: as for outcome 1
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 101 | 103 | 101
percentage of participants | 60.4 | 61.2 | 63.4

24. Secondary Outcome: PFS Per Modified RECIST Via Investigator Assessment in ITT Population
Description: PFS was defined as the time from randomization to the first occurrence of PD or death due to any cause. PD: at least a 20% increase in the sum of diameters of all target and new measurable lesions, taking as reference the smallest sum on study, including baseline, and an absolute increase of at least 5 mm. Kaplan-Meier methodology was used to estimate PFS.
Time Frame: as for outcome 1
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 101 | 103 | 101
months | 16.7 [11.4 to 22.6] | 10.9 [7.9 to 14.0] | 9.9 [8.1 to 14.1]
Statistical Analysis 1: Comparison: Atezolizumab and Bevacizumab vs Sunitinib; Test type: Superiority; p = 0.0863, Log Rank; Hazard Ratio (HR) = 0.72, 95% CI [0.50 to 1.05]
Statistical Analysis 2: Comparison: Atezolizumab vs Sunitinib; Test type: Superiority; p = 0.5922, Log Rank; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.77 to 1.57]

25. Secondary Outcome: Percentage of Participants With Disease Progression Per Modified RECIST Via Investigator Assessment or Death in IC1/2/3 Population
Description: as for outcome 23
Time Frame: as for outcome 1
Population: IC1/2/3 population
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 50 | 54 | 60
percentage of participants | 52.0 | 59.3 | 75.0

26. Secondary Outcome: PFS Per Modified RECIST Via Investigator Assessment in IC1/2/3 Population
Description: as for outcome 24
Time Frame: as for outcome 1
Population: IC1/2/3 population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 50 | 54 | 60
months | 21.7 [11.1 to NA] — Data could not be estimated due to high number of censored participants. | 10.9 [5.4 to 14.0] | 8.4 [5.8 to 11.3]
Statistical Analysis 1: Comparison: Atezolizumab and Bevacizumab vs Sunitinib; Test type: Superiority; p = 0.0021, Log Rank; Hazard Ratio (HR) = 0.43, 95% CI [0.25 to 0.75]
Statistical Analysis 2: Comparison: Atezolizumab vs Sunitinib; Test type: Superiority; p = 0.6566, Log Rank; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.56 to 1.44]

27. Secondary Outcome: Duration of Response (DOR) Per RECIST v1.1 Via IRC Assessment in ITT Population
Description: DOR was defined as the time from first observation of an objective response (CR or PR) until first observation of PD. CR: disappearance of all target and non-target lesions and (if applicable) normalization of tumor marker level; or reduction in short axis of any pathological lymph nodes (whether target or non-target) to <10 mm. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters; or persistence of one or more non-target lesion(s) and/or (if applicable) maintenance of tumor marker level above the normal limits. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline, and an absolute increase of at least 5 mm; appearance of one or more new target or non-target lesions; or unequivocal progression of existing non-target lesions. Kaplan-Meier methodology was used to estimate DOR.
Time Frame: From CR or PR until disease progression or death due to any cause (until data cut-off date 17 October 2016, up to approximately 2.75 years)
Population: ITT population. 'Overall Number of Participants Analyzed'=participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 32 | 26 | 29
months | 22.1 [19.4 to NA] — Data could not be estimated due to high number of censored participants. | NA [23.4 to NA] — Data could not be estimated due to high number of censored participants. | NA [NA to NA] — Data could not be estimated due to high number of censored participants.

28. Secondary Outcome: DOR Per RECIST v1.1 Via Investigator Assessment in ITT Population
Description: as for outcome 27
Time Frame: as for outcome 27
Population: ITT population. 'Overall Number of Participants Analyzed'=participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 35 | 24 | 33
months | NA [19.4 to NA] — Data could not be estimated due to high number of censored participants. | NA [NA to NA] — Data could not be estimated due to high number of censored participants. | 14.2 [13.0 to NA] — Data could not be estimated due to high number of censored participants.

29. Secondary Outcome: DOR Per RECIST v1.1 Via IRC Assessment in IC1/2/3 Population
Description: as for outcome 27
Time Frame: as for outcome 27
Population: IC1/2/3 population. 'Overall Number of Participants Analyzed'=participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 23 | 15 | 16
months | 22.1 [19.4 to NA] — Data could not be estimated due to high number of censored participants. | NA [23.4 to NA] — Data could not be estimated due to high number of censored participants. | NA [12.0 to NA] — Data could not be estimated due to high number of censored participants.

30. Secondary Outcome: DOR Per RECIST v1.1 Via Investigator Assessment in IC1/2/3 Population
Description: as for outcome 27
Time Frame: as for outcome 27
Population: IC1/2/3 population. 'Overall Number of Participants Analyzed'=participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 24 | 14 | 17
months | 22.4 [13.8 to NA] — Data could not be estimated due to high number of censored participants. | NA [NA to NA] — Data could not be estimated due to high number of censored participants. | 14.1 [11.1 to NA] — Data could not be estimated due to high number of censored participants.

31. Secondary Outcome: DOR Per Modified RECIST Via Investigator Assessment in ITT Population
Description: DOR was defined as the time from first observation of an objective response (CR or PR) until first observation of PD. CR: disappearance of all target and non-target lesions; or reduction in short axis of any pathological lymph nodes (whether target or non-target) to <10 mm. PR: at least a 30% decrease in the sum of diameters of target and all new measurable lesions, taking as reference the baseline sum of diameters, in absence of CR. PD: at least a 20% increase in the sum of diameters of all target and new measurable lesions, taking as reference the smallest sum on study, including baseline, and an absolute increase of at least 5 mm. Kaplan-Meier methodology was used to estimate DOR.
Time Frame: as for outcome 27
Population: ITT population. 'Overall Number of Participants Analyzed'=participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 38 | 26 | 34
months | NA [19.8 to NA] — Data could not be estimated due to high number of censored participants. | NA [NA to NA] — Data could not be estimated due to high number of censored participants. | 16.6 [13.6 to NA] — Data could not be estimated due to high number of censored participants.

32. Secondary Outcome: DOR Per Modified RECIST Via Investigator Assessment in IC1/2/3 Population
Description: as for outcome 31
Time Frame: as for outcome 27
Population: IC1/2/3 population. 'Overall Number of Participants Analyzed'=participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 26 | 15 | 18
months | 22.4 [19.4 to NA] — Data could not be estimated due to high number of censored participants. | NA [NA to NA] — Data could not be estimated due to high number of censored participants. | 16.6 [11.3 to NA] — Data could not be estimated due to high number of censored participants.

33. Secondary Outcome: Percentage of Participants Who Died in ITT Population
Time Frame: Randomization until death due to any cause (until data cut-off date 17 October 2016, up to approximately 2.75 years)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 101 | 103 | 101
percentage of participants | 38.6 | 35.0 | 30.7

34. Secondary Outcome: Overall Survival (OS) in ITT Population
Description: OS was defined as the time from the date of randomization to the date of death due to any cause. Kaplan-Meier methodology was used to estimate OS.
Time Frame: Randomization until death due to any cause (until data cut-off date 17 October 2016, up to approximately 2.75 years)
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 101 | 103 | 101
months | NA [23.9 to NA] — Data could not be estimated due to high number of censored participants. | NA [30.2 to NA] — Data could not be estimated due to high number of censored participants. | NA [27.2 to NA] — Data could not be estimated due to high number of censored participants.
Statistical Analysis 1: Comparison: Atezolizumab and Bevacizumab vs Sunitinib; Test type: Superiority; p = 0.2867, Log Rank; Hazard Ratio (HR) = 1.30, 95% CI 2-sided [0.80 to 2.13]
Statistical Analysis 2: Comparison: Atezolizumab vs Sunitinib; Test type: Superiority; p = 0.8039, Log Rank; Hazard Ratio (HR) = 1.06, 95% CI [0.65 to 1.73]

35. Secondary Outcome: Percentage of Participants Who Died in IC1/2/3 Population
Time Frame: Randomization until death due to any cause (until data cut-off date 17 October 2016, up to approximately 2.75 years)
Population: IC1/2/3 population
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 50 | 54 | 60
percentage of participants | 38.0 | 39.8 | 35.0

36. Secondary Outcome: OS in IC1/2/3 Population
Description: as for outcome 34
Time Frame: Randomization until death due to any cause (until data cut-off date 17 October 2016, up to approximately 2.75 years)
Population: IC1/2/3 population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 50 | 54 | 60
months | 27.3 [24.6 to NA] — Data could not be estimated due to high number of censored participants. | 30.2 [23.3 to NA] — Data could not be estimated due to high number of censored participants. | NA [22.4 to NA] — Data could not be estimated due to high number of censored participants.
Statistical Analysis 1: Comparison: Atezolizumab and Bevacizumab vs Sunitinib; Test type: Superiority; p = 0.7879, Log Rank; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.47 to 1.78]
Statistical Analysis 2: Comparison: Atezolizumab vs Sunitinib; Test type: Superiority; p = 0.9065, Log Rank; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.52 to 1.80]

37. Secondary Outcome: Percentage of Participants With Objective Response Per RECIST v1.1 Via Investigator Assessment in Crossover Population
Description: as for outcome 18
Time Frame: From start of crossover treatment until disease progression or death due to any cause (until data cut-off date 17 October 2016, up to approximately 2.75 years)
Population: Crossover population included participants in atezolizumab or sunitinib arms who had crossed over to the atezolizumab and bevacizumab arm. 'Overall Number of Participants Analyzed'=participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Atezolizumab (Crossover): Among the participants assigned to atezolizumab initially, those participants who upon disease progression, crossed over to receive atezolizumab and bevacizumab combination until disease progression, lack of clinical benefit, unacceptable toxicity, withdrawal from study, or study completion or termination, were included in this group. Atezolizumab 1200 mg and bevacizumab 15 mg/kg were administered as IV infusions q3w on Day 1 and Day 22 of each 6-week cycle.
- Sunitinib (Crossover): Among the participants assigned to sunitinib initially, those participants who upon disease progression, crossed over to receive atezolizumab and bevacizumab combination until disease progression, lack of clinical benefit, unacceptable toxicity, withdrawal from study, or study completion or termination, were included in this group. Atezolizumab 1200 mg and bevacizumab 15 mg/kg were administered as IV infusions q3w on Day 1 and Day 22 of each 6-week cycle.
Arm/Group | Atezolizumab (Crossover) | Sunitinib (Crossover)
Number analyzed (Participants) | 41 | 54
percentage of participants | 24.4 [12.36 to 40.30] | 27.8 [16.46 to 41.64]

38. Secondary Outcome: DOR Per RECIST v1.1 Via Investigator Assessment in Crossover Population
Description: as for outcome 27
Time Frame: as for outcome 37
Population: Crossover population. 'Overall Number of Participants Analyzed'=participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab (Crossover) | Sunitinib (Crossover)
Number analyzed (Participants) | 10 | 15
months | NA [7.2 to NA] — Data could not be estimated due to high number of censored participants. | NA [11.1 to NA] — Data could not be estimated due to high number of censored participants.

39. Secondary Outcome: Percentage of Participants With Disease Progression Per RECIST v1.1 Via Investigator Assessment or Death in Crossover Population
Description: as for outcome 3
Time Frame: as for outcome 37
Population: Crossover population
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab (Crossover) | Sunitinib (Crossover)
Number analyzed (Participants) | 44 | 57
percentage of participants | 59.1 | 68.4

40. Secondary Outcome: PFS Per RECIST v.1.1 Via Investigator Assessment in Crossover Population
Description: as for outcome 2
Time Frame: as for outcome 37
Population: Crossover population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab (Crossover) | Sunitinib (Crossover)
Number analyzed (Participants) | 44 | 57
months | 12.6 [6.0 to 17.7] | 8.3 [3.1 to 11.2]

41. Secondary Outcome: Percentage of Participants With Anti-Therapeutic Antibodies (ATA) to Atezolizumab
Description: This outcome measure was planned to be analyzed in 'Atezolizumab' and 'Atezolizumab and Bevacizumab' arms only.
Time Frame: Cycle 1 Day 1 until treatment discontinuation (until data cut-off date 17 October 2016, up to approximately 2.75 years) (1 cycle=6 weeks)
Population: ATA evaluable population included participants at baseline who had a baseline ATA sample and post-baseline participants who had at least one ATA sample and had received at least one dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab
Number analyzed (Participants) | 97 | 96
percentage of participants | 34.0 | 25.0

42. Secondary Outcome: Maximum Serum Concentration (Cmax) of Atezolizumab
Time Frame: 30 minutes after end of infusion on Cycle 1 Day 1 (1 cycle=6 weeks) (infusion length for first dose=60 minutes)
Population: The pharmacokinetic (PK) evaluable population included participants who received at least one dose of study drug and had sufficient PK sample collected within the time specified in the protocol. 'Overall Number of Participants Analyzed'=participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Atezolizumab (Crossover) | Sunitinib (Crossover)
Number analyzed (Participants) | 95 | 93 | 41 | 53
micrograms per milliliter (mcg/mL) | 335 (86.0) | 358 (93.1) | 418 (114) | 314 (87.1)

43. Secondary Outcome: Minimum Serum Concentration (Cmin) of Atezolizumab
Time Frame: Pre-infusion (0 hour) on Day 1 of Cycles 2 and 4; Day 22 of Cycles 1, 2, and 4 (1 cycle=6 weeks) (infusion length=30-60 minutes)
Population: PK evaluable population. 'Overall Number of Participants Analyzed'=participants evaluable for this outcome measure. 'Number Analyzed'=participants evaluable for this outcome measure at specified timepoint for each arm respectively.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Atezolizumab (Crossover) | Sunitinib (Crossover)
Number analyzed (Participants) | 98 | 94 | 42 | 52
mcg/mL
  Cycle 1 Day 22 | 72.6 (29.5) | 79.9 (26.1) | 174 (121) | 73.2 (31.5)
  Cycle 2 Day 1: number analyzed (Participants) | 89 | 88 | 38 | 49
  Cycle 2 Day 1 | 122 (50.4) | 125 (47.4) | 158 (101) | 106 (45.2)
  Cycle 2 Day 22: number analyzed (Participants) | 85 | 88 | 38 | 44
  Cycle 2 Day 22 | 152 (65.3) | 159 (84.6) | 164 (70.7) | 141 (85.5)
  Cycle 4 Day 1: number analyzed (Participants) | 79 | 66 | 28 | 34
  Cycle 4 Day 1 | 183 (90.5) | 192 (77.6) | 154 (62.7) | 174 (75.7)
  Cycle 4 Day 22: number analyzed (Participants) | 71 | 65 | 25 | 29
  Cycle 4 Day 22 | 190 (86.3) | 200 (90.0) | 163 (70.5) | 172 (78.8)

44. Secondary Outcome: Cmax of Bevacizumab
Time Frame: 30 minutes after end of infusion on Day 1 of Cycles 1 and 2 (1 cycle=6 weeks) (infusion length=30-90 minutes)
Population: PK evaluable population. 'Overall Number of Participants Analyzed'=participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab (Crossover) | Sunitinib (Crossover)
Number analyzed (Participants) | 86 | 34 | 44
mcg/mL | 89.8 (39.4) | 433 (115) | 455 (106)

45. Secondary Outcome: Cmin of Bevacizumab
Time Frame: For Atezolizumab and Bevacizumab Arm: at First-line treatment discontinuation (up to approximately 2.75 years); For Crossover Arms: pre-infusion (0 hour) on Day 1 of Cycle 2 (1 cycle=6 weeks) (infusion length=30-90 minutes)
Population: PK evaluable population. 'Overall Number of Participants Analyzed'=participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab (Crossover) | Sunitinib (Crossover)
Number analyzed (Participants) | 42 | 39 | 42
mcg/mL | 75.2 (72.1) | 101 (48.7) | 95.9 (43.9)

46. Secondary Outcome: M.D. Anderson Symptom Inventory (MDASI) Interference Score
Description: MDASI questionnaire comprises of 2 parts: symptoms (16 items), interference with daily life (6 items). Participants were asked to rate how much their symptoms interfered with general activity, mood, work, relations with other people, walking, and enjoyment of life during the last 24 hours. Each item in the interference score was answered on a scale of 0 (did not interfere) to 10 (interfered completely). The mean score of all 6 items was reported on the scale of 0 (did not interfere) to 10 (interfered completely).
Time Frame: Days 1 and 22 of Cycles 1 to 24; Day 1 of Cycle 25; treatment discontinuation (up to approximately 2.75 years) (1 cycle=6 weeks)
Population: Patient Reported Outcome (PRO)-evaluable population: randomized participants who had non-missing baseline assessment and at least 1 post-baseline assessment. 'Overall Number of Participants Analyzed'=participants evaluable for this outcome. 'Number Analyzed'=participants evaluable for this outcome at specified timepoint for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 96 | 95 | 93
units on a scale
  Cycle 1 Day 1 | 1.60 (1.97) | 1.38 (2.03) | 1.79 (2.39)
  Cycle 1 Day 22: number analyzed (Participants) | 93 | 88 | 88
  Cycle 1 Day 22 | 2.08 (2.34) | 1.26 (2.07) | 3.16 (2.65)
  Cycle 2 Day 1: number analyzed (Participants) | 86 | 82 | 80
  Cycle 2 Day 1 | 1.56 (1.82) | 1.20 (1.72) | 1.83 (2.19)
  Cycle 2 Day 22: number analyzed (Participants) | 82 | 80 | 77
  Cycle 2 Day 22 | 1.57 (1.83) | 1.04 (1.62) | 2.50 (2.47)
  Cycle 3 Day 1: number analyzed (Participants) | 77 | 65 | 69
  Cycle 3 Day 1 | 1.72 (2.15) | 0.90 (1.43) | 1.49 (2.01)
  Cycle 3 Day 22: number analyzed (Participants) | 74 | 63 | 63
  Cycle 3 Day 22 | 1.66 (2.07) | 1.01 (1.58) | 2.20 (2.42)
  Cycle 4 Day 1: number analyzed (Participants) | 72 | 61 | 62
  Cycle 4 Day 1 | 1.59 (2.11) | 1.24 (1.99) | 1.61 (2.24)
  Cycle 4 Day 22: number analyzed (Participants) | 68 | 61 | 59
  Cycle 4 Day 22 | 1.68 (2.31) | 1.26 (1.98) | 1.92 (2.00)
  Cycle 5 Day 1: number analyzed (Participants) | 60 | 52 | 53
  Cycle 5 Day 1 | 1.70 (2.29) | 0.69 (1.11) | 1.53 (1.96)
  Cycle 5 Day 22: number analyzed (Participants) | 60 | 50 | 47
  Cycle 5 Day 22 | 1.80 (2.29) | 0.67 (1.33) | 1.97 (2.21)
  Cycle 6 Day 1: number analyzed (Participants) | 57 | 47 | 49
  Cycle 6 Day 1 | 1.91 (2.54) | 0.64 (1.13) | 1.39 (1.76)
  Cycle 6 Day 22: number analyzed (Participants) | 56 | 49 | 44
  Cycle 6 Day 22 | 1.80 (2.38) | 0.63 (1.12) | 2.00 (2.23)
  Cycle 7 Day 1: number analyzed (Participants) | 51 | 41 | 41
  Cycle 7 Day 1 | 1.99 (2.49) | 0.53 (0.78) | 1.00 (1.09)
  Cycle 7 Day 22: number analyzed (Participants) | 51 | 40 | 38
  Cycle 7 Day 22 | 2.01 (2.45) | 0.59 (0.93) | 1.15 (1.04)
  Cycle 8 Day 1: number analyzed (Participants) | 50 | 41 | 39
  Cycle 8 Day 1 | 1.88 (2.26) | 0.55 (0.85) | 0.94 (1.04)
  Cycle 8 Day 22: number analyzed (Participants) | 51 | 38 | 36
  Cycle 8 Day 22 | 1.81 (2.41) | 0.58 (0.91) | 1.34 (1.39)
  Cycle 9 Day 1: number analyzed (Participants) | 46 | 34 | 33
  Cycle 9 Day 1 | 1.75 (2.24) | 0.55 (0.90) | 1.16 (1.22)
  Cycle 9 Day 22: number analyzed (Participants) | 46 | 32 | 28
  Cycle 9 Day 22 | 1.64 (2.16) | 0.58 (0.89) | 1.57 (1.61)
  Cycle 10 Day 1: number analyzed (Participants) | 45 | 33 | 28
  Cycle 10 Day 1 | 1.43 (1.82) | 0.81 (1.13) | 1.08 (1.40)
  Cycle 10 Day 22: number analyzed (Participants) | 43 | 33 | 29
  Cycle 10 Day 22 | 1.55 (2.09) | 0.70 (1.10) | 1.49 (1.78)
  Cycle 11 Day 1: number analyzed (Participants) | 41 | 30 | 29
  Cycle 11 Day 1 | 1.65 (2.13) | 0.61 (0.95) | 0.98 (1.00)
  Cycle 11 Day 22: number analyzed (Participants) | 38 | 28 | 26
  Cycle 11 Day 22 | 1.35 (1.81) | 0.78 (1.07) | 1.47 (1.61)
  Cycle 12 Day 1: number analyzed (Participants) | 39 | 28 | 29
  Cycle 12 Day 1 | 1.21 (1.69) | 0.68 (1.15) | 0.84 (0.83)
  Cycle 12 Day 22: number analyzed (Participants) | 38 | 25 | 26
  Cycle 12 Day 22 | 1.51 (2.23) | 0.53 (0.99) | 1.41 (1.53)
  Cycle 13 Day 1: number analyzed (Participants) | 35 | 23 | 24
  Cycle 13 Day 1 | 1.50 (2.16) | 0.68 (1.07) | 1.26 (1.45)
  Cycle 13 Day 22: number analyzed (Participants) | 37 | 23 | 20
  Cycle 13 Day 22 | 1.45 (2.32) | 0.67 (1.10) | 1.32 (1.37)
  Cycle 14 Day 1: number analyzed (Participants) | 35 | 21 | 23
  Cycle 14 Day 1 | 1.60 (2.24) | 0.67 (0.95) | 1.07 (1.31)
  Cycle 14 Day 22: number analyzed (Participants) | 35 | 19 | 20
  Cycle 14 Day 22 | 1.40 (2.09) | 0.63 (0.94) | 1.50 (1.48)
  Cycle 15 Day 1: number analyzed (Participants) | 31 | 17 | 21
  Cycle 15 Day 1 | 1.16 (1.74) | 0.84 (1.16) | 1.50 (1.64)
  Cycle 15 Day 22: number analyzed (Participants) | 28 | 13 | 15
  Cycle 15 Day 22 | 1.48 (1.92) | 0.71 (1.10) | 2.08 (1.64)
  Cycle 16 Day 1: number analyzed (Participants) | 25 | 13 | 14
  Cycle 16 Day 1 | 0.87 (0.99) | 0.85 (1.40) | 1.07 (1.22)
  Cycle 16 Day 22: number analyzed (Participants) | 23 | 9 | 14
  Cycle 16 Day 22 | 0.72 (0.93) | 0.87 (1.30) | 2.04 (2.24)
  Cycle 17 Day 1: number analyzed (Participants) | 18 | 10 | 8
  Cycle 17 Day 1 | 0.98 (0.99) | 0.57 (0.75) | 0.71 (0.95)
  Cycle 17 Day 22: number analyzed (Participants) | 14 | 8 | 8
  Cycle 17 Day 22 | 0.73 (1.02) | 0.65 (0.97) | 1.21 (1.32)
  Cycle 18 Day 1: number analyzed (Participants) | 12 | 8 | 7
  Cycle 18 Day 1 | 0.93 (1.07) | 0.71 (0.98) | 0.95 (1.15)
  Cycle 18 Day 22: number analyzed (Participants) | 13 | 6 | 7
  Cycle 18 Day 22 | 0.79 (1.06) | 0.33 (0.41) | 1.05 (1.42)
  Cycle 19 Day 1: number analyzed (Participants) | 11 | 6 | 7
  Cycle 19 Day 1 | 1.11 (1.25) | 0.31 (0.34) | 1.33 (1.66)
  Cycle 19 Day 22: number analyzed (Participants) | 10 | 5 | 7
  Cycle 19 Day 22 | 0.97 (1.37) | 0.30 (0.41) | 1.55 (1.69)
  Cycle 20 Day 1: number analyzed (Participants) | 8 | 4 | 5
  Cycle 20 Day 1 | 1.19 (1.31) | 0.21 (0.42) | 0.90 (1.07)
  Cycle 20 Day 22: number analyzed (Participants) | 5 | 4 | 4
  Cycle 20 Day 22 | 1.10 (1.30) | 0.04 (0.08) | 1.67 (1.56)
  Cycle 21 Day 1: number analyzed (Participants) | 5 | 2 | 3
  Cycle 21 Day 1 | 1.17 (1.42) | 0.00 (0.00) | 0.78 (1.07)
  Cycle 21 Day 22: number analyzed (Participants) | 5 | 1 | 2
  Cycle 21 Day 22 | 1.23 (1.51) | 0.00 (NA) — Standard deviation was not estimable for single evaluable participant. | 1.25 (1.53)
  Cycle 22 Day 1: number analyzed (Participants) | 4 | 1 | 2
  Cycle 22 Day 1 | 0.54 (0.76) | 0.00 (NA) — Standard deviation was not estimable for single evaluable participant. | 0.83 (0.71)
  Cycle 22 Day 22: number analyzed (Participants) | 3 | 1 | 2
  Cycle 22 Day 22 | 0.94 (1.07) | 0.00 (NA) — Standard deviation was not estimable for single evaluable participant. | 1.25 (1.53)
  Cycle 23 Day 1: number analyzed (Participants) | 2 | 1 | 2
  Cycle 23 Day 1 | 1.67 (1.89) | 0.00 (NA) — Standard deviation was not estimable for single evaluable participant. | 1.58 (2.00)
  Cycle 23 Day 22: number analyzed (Participants) | 2 | 1 | 2
  Cycle 23 Day 22 | 1.25 (1.77) | 0.00 (NA) — Standard deviation was not estimable for single evaluable participant. | 2.67 (2.36)
  Cycle 24 Day 1: number analyzed (Participants) | 1 | 1 | 1
  Cycle 24 Day 1 | 2.33 (NA) — Standard deviation was not estimable for single evaluable participant. | 0.00 (NA) — Standard deviation was not estimable for single evaluable participant. | 1.67 (NA) — Standard deviation was not estimable for single evaluable participant.
  Cycle 24 Day 22: number analyzed (Participants) | 0 | 1 | 1
  Cycle 24 Day 22 |  | 0.00 (NA) — Standard deviation was not estimable for single evaluable participant. | 0.50 (NA) — Standard deviation was not estimable for single evaluable participant.
  Cycle 25 Day 1: number analyzed (Participants) | 0 | 1 | 0
  Cycle 25 Day 1 |  | 0.00 (NA) — Standard deviation was not estimable for single evaluable participant. |
  Treatment discontinuation: number analyzed (Participants) | 46 | 39 | 39
  Treatment discontinuation | 2.54 (2.66) | 2.29 (2.54) | 3.49 (3.16)

47. Secondary Outcome: Brief Fatigue Inventory (BFI) Fatigue Level Score
Description: BFI questionnaire comprises of 2 parts: fatigue level (3 items), interference with daily life (1 item with 6 sub-items). Each items in the fatigue level score was answered on a scale of 0 (no fatigue) to 10 (as bad as you can imagine). The mean score of all 3 items was reported on the scale of 0 (no fatigue) to 10 (as bad as you can imagine).
Time Frame: as for outcome 46
Population: PRO-evaluable population. 'Overall Number of Participants Analyzed'=participants evaluable for this outcome measure. 'Number Analyzed'=participants evaluable for this outcome measure at specified timepoint for each arm respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 95 | 94 | 93
units on a scale
  Cycle 1 Day 1: number analyzed (Participants) | 93 | 93 | 92
  Cycle 1 Day 1 | 2.80 (2.64) | 2.52 (2.72) | 2.66 (2.74)
  Cycle 1 Day 22: number analyzed (Participants) | 90 | 86 | 89
  Cycle 1 Day 22 | 3.80 (2.86) | 2.55 (2.60) | 4.42 (3.09)
  Cycle 2 Day 1: number analyzed (Participants) | 86 | 79 | 79
  Cycle 2 Day 1 | 3.21 (2.61) | 2.63 (2.69) | 2.86 (2.76)
  Cycle 2 Day 22: number analyzed (Participants) | 81 | 82 | 78
  Cycle 2 Day 22 | 3.15 (2.61) | 2.57 (2.74) | 3.69 (2.74)
  Cycle 3 Day 1: number analyzed (Participants) | 76 | 64 | 69
  Cycle 3 Day 1 | 2.91 (2.60) | 2.11 (2.42) | 2.35 (2.44)
  Cycle 3 Day 22: number analyzed (Participants) | 74 | 62 | 63
  Cycle 3 Day 22 | 2.93 (2.67) | 2.31 (2.71) | 3.60 (3.09)
  Cycle 4 Day 1: number analyzed (Participants) | 72 | 62 | 62
  Cycle 4 Day 1 | 3.21 (2.66) | 2.32 (2.86) | 2.39 (2.47)
  Cycle 4 Day 22: number analyzed (Participants) | 66 | 61 | 59
  Cycle 4 Day 22 | 3.06 (2.68) | 2.33 (2.94) | 3.15 (2.57)
  Cycle 5 Day 1: number analyzed (Participants) | 59 | 51 | 53
  Cycle 5 Day 1 | 2.97 (2.83) | 1.59 (2.03) | 2.32 (2.62)
  Cycle 5 Day 22: number analyzed (Participants) | 60 | 50 | 47
  Cycle 5 Day 22 | 3.02 (2.87) | 1.34 (1.81) | 2.91 (2.86)
  Cycle 6 Day 1: number analyzed (Participants) | 57 | 48 | 49
  Cycle 6 Day 1 | 3.05 (2.83) | 1.42 (1.90) | 2.22 (2.48)
  Cycle 6 Day 22: number analyzed (Participants) | 56 | 49 | 44
  Cycle 6 Day 22 | 3.23 (2.94) | 1.39 (2.01) | 3.09 (2.69)
  Cycle 7 Day 1: number analyzed (Participants) | 51 | 40 | 40
  Cycle 7 Day 1 | 3.16 (2.81) | 1.33 (1.91) | 1.68 (1.75)
  Cycle 7 Day 22: number analyzed (Participants) | 51 | 41 | 38
  Cycle 7 Day 22 | 2.86 (2.60) | 1.24 (1.67) | 2.16 (1.87)
  Cycle 8 Day 1: number analyzed (Participants) | 50 | 41 | 39
  Cycle 8 Day 1 | 2.80 (2.56) | 1.12 (1.68) | 1.72 (1.70)
  Cycle 8 Day 22: number analyzed (Participants) | 51 | 38 | 36
  Cycle 8 Day 22 | 2.88 (2.80) | 1.24 (1.75) | 2.58 (2.13)
  Cycle 9 Day 1: number analyzed (Participants) | 46 | 35 | 34
  Cycle 9 Day 1 | 3.09 (2.81) | 1.11 (1.55) | 2.12 (2.48)
  Cycle 9 Day 22: number analyzed (Participants) | 46 | 32 | 28
  Cycle 9 Day 22 | 2.80 (2.73) | 1.19 (1.71) | 2.64 (2.57)
  Cycle 10 Day 1: number analyzed (Participants) | 45 | 34 | 28
  Cycle 10 Day 1 | 2.80 (2.58) | 1.29 (1.88) | 2.11 (2.23)
  Cycle 10 Day 22: number analyzed (Participants) | 43 | 33 | 29
  Cycle 10 Day 22 | 2.91 (2.83) | 1.33 (1.90) | 2.24 (2.43)
  Cycle 11 Day 1: number analyzed (Participants) | 40 | 30 | 28
  Cycle 11 Day 1 | 2.98 (2.71) | 1.40 (1.96) | 1.93 (1.65)
  Cycle 11 Day 22: number analyzed (Participants) | 37 | 29 | 26
  Cycle 11 Day 22 | 2.59 (2.44) | 1.72 (2.23) | 2.42 (2.12)
  Cycle 12 Day 1: number analyzed (Participants) | 39 | 28 | 29
  Cycle 12 Day 1 | 2.31 (2.25) | 1.25 (1.96) | 1.66 (1.67)
  Cycle 12 Day 22: number analyzed (Participants) | 38 | 25 | 26
  Cycle 12 Day 22 | 2.79 (2.46) | 1.44 (2.12) | 2.27 (2.05)
  Cycle 13 Day 1: number analyzed (Participants) | 36 | 23 | 24
  Cycle 13 Day 1 | 2.69 (2.57) | 1.65 (2.17) | 2.08 (1.56)
  Cycle 13 Day 22: number analyzed (Participants) | 37 | 22 | 20
  Cycle 13 Day 22 | 2.97 (2.97) | 1.55 (2.13) | 2.60 (2.28)
  Cycle 14 Day 1: number analyzed (Participants) | 35 | 20 | 23
  Cycle 14 Day 1 | 2.94 (2.94) | 1.45 (2.14) | 2.30 (2.34)
  Cycle 14 Day 22: number analyzed (Participants) | 35 | 18 | 20
  Cycle 14 Day 22 | 2.83 (2.85) | 1.61 (2.00) | 2.60 (2.09)
  Cycle 15 Day 1: number analyzed (Participants) | 30 | 17 | 20
  Cycle 15 Day 1 | 2.73 (2.56) | 1.76 (2.19) | 2.60 (2.33)
  Cycle 15 Day 22: number analyzed (Participants) | 28 | 13 | 16
  Cycle 15 Day 22 | 2.61 (2.79) | 0.92 (1.12) | 2.94 (1.61)
  Cycle 16 Day 1: number analyzed (Participants) | 25 | 13 | 14
  Cycle 16 Day 1 | 1.88 (1.99) | 1.54 (2.07) | 2.21 (2.42)
  Cycle 16 Day 22: number analyzed (Participants) | 23 | 9 | 13
  Cycle 16 Day 22 | 1.70 (1.61) | 2.11 (2.15) | 2.85 (2.19)
  Cycle 17 Day 1: number analyzed (Participants) | 18 | 10 | 8
  Cycle 17 Day 1 | 1.78 (1.59) | 1.60 (1.96) | 1.50 (1.51)
  Cycle 17 Day 22: number analyzed (Participants) | 14 | 8 | 8
  Cycle 17 Day 22 | 2.00 (1.80) | 2.13 (2.42) | 2.38 (1.60)
  Cycle 18 Day 1: number analyzed (Participants) | 13 | 8 | 7
  Cycle 18 Day 1 | 2.23 (1.74) | 1.88 (2.23) | 1.71 (1.70)
  Cycle 18 Day 22: number analyzed (Participants) | 13 | 6 | 7
  Cycle 18 Day 22 | 1.92 (2.14) | 1.67 (2.07) | 2.14 (2.19)
  Cycle 19 Day 1: number analyzed (Participants) | 12 | 6 | 7
  Cycle 19 Day 1 | 2.17 (2.48) | 1.50 (1.97) | 2.29 (3.30)
  Cycle 19 Day 22: number analyzed (Participants) | 10 | 5 | 7
  Cycle 19 Day 22 | 1.90 (2.42) | 1.40 (2.19) | 3.29 (2.43)
  Cycle 20 Day 1: number analyzed (Participants) | 8 | 4 | 5
  Cycle 20 Day 1 | 3.00 (3.16) | 1.25 (2.50) | 1.80 (1.30)
  Cycle 20 Day 22: number analyzed (Participants) | 5 | 4 | 4
  Cycle 20 Day 22 | 2.40 (3.05) | 1.50 (3.00) | 2.25 (2.06)
  Cycle 21 Day 1: number analyzed (Participants) | 5 | 2 | 3
  Cycle 21 Day 1 | 2.60 (2.97) | 2.50 (3.54) | 1.67 (1.53)
  Cycle 21 Day 22: number analyzed (Participants) | 5 | 1 | 2
  Cycle 21 Day 22 | 2.40 (1.95) | 0.00 (NA) — Standard deviation was not estimable for single evaluable participant. | 2.00 (1.41)
  Cycle 22 Day 1: number analyzed (Participants) | 4 | 1 | 2
  Cycle 22 Day 1 | 1.25 (1.89) | 0.00 (NA) — Standard deviation was not estimable for single evaluable participant. | 2.00 (1.41)
  Cycle 22 Day 22: number analyzed (Participants) | 3 | 1 | 2
  Cycle 22 Day 22 | 1.33 (2.31) | 0.00 (NA) — Standard deviation was not estimable for single evaluable participant. | 3.00 (2.83)
  Cycle 23 Day 1: number analyzed (Participants) | 2 | 1 | 2
  Cycle 23 Day 1 | 2.50 (3.54) | 0.00 (NA) — Standard deviation was not estimable for single evaluable participant. | 2.00 (2.83)
  Cycle 23 Day 22: number analyzed (Participants) | 2 | 1 | 2
  Cycle 23 Day 22 | 2.00 (2.83) | 0.00 (NA) — Standard deviation was not estimable for single evaluable participant. | 4.50 (3.54)
  Cycle 24 Day 1: number analyzed (Participants) | 1 | 1 | 1
  Cycle 24 Day 1 | 4.00 (NA) — Standard deviation was not estimable for single evaluable participant. | 0.00 (NA) — Standard deviation was not estimable for single evaluable participant. | 2.00 (NA) — Standard deviation was not estimable for single evaluable participant.
  Cycle 24 Day 22: number analyzed (Participants) | 0 | 1 | 1
  Cycle 24 Day 22 |  | 0.00 (NA) — Standard deviation was not estimable for single evaluable participant. | 0.00 (NA) — Standard deviation was not estimable for single evaluable participant.
  Cycle 25 Day 1: number analyzed (Participants) | 0 | 1 | 0
  Cycle 25 Day 1 |  | 0.00 (NA) — Standard deviation was not estimable for single evaluable participant. |
  Treatment discontinuation: number analyzed (Participants) | 46 | 39 | 40
  Treatment discontinuation | 3.74 (2.82) | 3.95 (3.27) | 3.75 (3.09)

48. Other Pre Specified Outcome: EuroQoL 5 Dimension (EQ-5D) Questionnaire Score
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state. Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: as for outcome 46
Population: As this outcome was pre-specified as an exploratory outcome, no results are reported.
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 60 months.
Description: Safety-evaluable population included all participants who received at least one dose of any study medication. Adverse events were reported separately for crossed over participants.
Arm/Group | Atezolizumab and Bevacizumab | Atezolizumab | Sunitinib | Atezolizumab (Crossover) | Sunitinib (Crossover)
Serious Adverse Events (participants affected / at risk) | 49/101 | 37/103 | 28/100 | 15/46 | 22/63
Other Adverse Events (participants affected / at risk) | 99/101 | 94/103 | 99/100 | 44/46 | 57/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atezolizumab and Bevacizumab (N=101) | Atezolizumab (N=103) | Sunitinib (N=100) | Atezolizumab (Crossover) (N=46) | Sunitinib (Crossover) (N=63)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 2
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Autoimmune pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 2 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3
Pancreatic fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 2
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 1 | 1
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 1
Pain (General disorders) | 1 | 0 | 1 | 0 | 3
Pyrexia (General disorders) | 2 | 4 | 2 | 0 | 2
Sudden death (General disorders) | 0 | 0 | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Chest wall abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 3 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 3 | 0 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pancreatic abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 2 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Spinal cord infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 2 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Autoimmune neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Demyelination (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Nerve root compression (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 3 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 3 | 2 | 1 | 2 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 2 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 0
Laryngeal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Limb Operation (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 4 | 0 | 2 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Colitis microscopic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 1 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Biliary sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Psoas abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Asparate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Intracranial haematoma (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Paresis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atezolizumab and Bevacizumab (N=101) | Atezolizumab (N=103) | Sunitinib (N=100) | Atezolizumab (Crossover) (N=46) | Sunitinib (Crossover) (N=63)
Anaemia (Blood and lymphatic system disorders) | 11 | 19 | 18 | 2 | 9
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 9 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 12 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 1 | 15 | 2 | 4
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 3 | 0
Hypothyroidism (Endocrine disorders) | 19 | 12 | 20 | 8 | 7
Abdominal distension (Gastrointestinal disorders) | 8 | 2 | 3 | 5 | 7
Abdominal pain (Gastrointestinal disorders) | 17 | 8 | 16 | 10 | 15
Abdominal pain upper (Gastrointestinal disorders) | 4 | 2 | 9 | 0 | 0
Constipation (Gastrointestinal disorders) | 30 | 16 | 30 | 9 | 14
Diarrhoea (Gastrointestinal disorders) | 36 | 20 | 62 | 13 | 19
Dry mouth (Gastrointestinal disorders) | 12 | 12 | 9 | 5 | 5
Dyspepsia (Gastrointestinal disorders) | 8 | 4 | 20 | 3 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 | 3 | 13 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 7 | 0 | 1 | 3 | 2
Nausea (Gastrointestinal disorders) | 40 | 19 | 46 | 14 | 21
Oral pain (Gastrointestinal disorders) | 4 | 0 | 7 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 15 | 3 | 25 | 6 | 5
Vomiting (Gastrointestinal disorders) | 20 | 8 | 21 | 6 | 16
Asthenia (General disorders) | 7 | 8 | 7 | 1 | 7
Chest pain (General disorders) | 7 | 5 | 6 | 4 | 1
Chills (General disorders) | 5 | 8 | 13 | 0 | 0
Fatigue (General disorders) | 62 | 52 | 70 | 19 | 27
Influenza like illness (General disorders) | 8 | 6 | 3 | 0 | 0
Mucosal inflammation (General disorders) | 18 | 4 | 33 | 6 | 4
Oedema peripheral (General disorders) | 20 | 12 | 10 | 8 | 10
Pain (General disorders) | 16 | 7 | 10 | 0 | 0
Pyrexia (General disorders) | 19 | 23 | 10 | 6 | 10
Nasopharyngitis (Infections and infestations) | 11 | 8 | 2 | 0 | 0
Rhinitis (Infections and infestations) | 8 | 6 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 15 | 5 | 3 | 4 | 4
Upper respiratory tract infection (Infections and infestations) | 14 | 11 | 5 | 8 | 2
Urinary tract infection (Infections and infestations) | 10 | 8 | 3 | 1 | 4
Alanine aminotransferase increased (Investigations) | 14 | 7 | 15 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 10 | 7 | 17 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 8 | 3 | 6 | 0 | 0
Blood creatinine increased (Investigations) | 13 | 17 | 14 | 10 | 8
Platelet count decreased (Investigations) | 2 | 2 | 6 | 3 | 0
Weight decreased (Investigations) | 18 | 5 | 10 | 2 | 6
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 3 | 3
Protein total increased (Investigations) | 0 | 0 | 0 | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 23 | 11 | 30 | 4 | 15
Dehydration (Metabolism and nutrition disorders) | 11 | 5 | 4 | 3 | 6
Hypercalcaemia (Metabolism and nutrition disorders) | 10 | 4 | 4 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 13 | 5 | 5 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 15 | 6 | 6 | 4 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 | 2 | 5 | 3 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 | 2 | 6 | 2 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 12 | 5 | 7 | 5 | 10
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 11 | 11 | 4 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 40 | 19 | 19 | 17 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 19 | 18 | 20 | 8 | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 2 | 6 | 4 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 22 | 10 | 6 | 9 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 10 | 15 | 3 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 10 | 5 | 8 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 | 8 | 17 | 9 | 6
Dizziness (Nervous system disorders) | 13 | 9 | 13 | 4 | 6
Dysgeusia (Nervous system disorders) | 12 | 3 | 30 | 0 | 0
Headache (Nervous system disorders) | 35 | 16 | 23 | 7 | 13
Neuropathy peripheral (Nervous system disorders) | 5 | 1 | 5 | 0 | 0
Paraesthesia (Nervous system disorders) | 8 | 8 | 11 | 1 | 4
Depression (Psychiatric disorders) | 9 | 5 | 7 | 2 | 4
Insomnia (Psychiatric disorders) | 10 | 7 | 12 | 3 | 8
Dysuria (Renal and urinary disorders) | 1 | 7 | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 3 | 10 | 9 | 4 | 4
Proteinuria (Renal and urinary disorders) | 38 | 10 | 9 | 21 | 25
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 2
Nocturia (Renal and urinary disorders) | 6 | 2 | 4 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 26 | 25 | 14 | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 18 | 2 | 4 | 9 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 18 | 18 | 8 | 10
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 8 | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 29 | 2 | 12 | 13 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12 | 11 | 3 | 5 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 11 | 3 | 6 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 5 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 3 | 3 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 13 | 15 | 10 | 5 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 8 | 5 | 7 | 4 | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 0 | 41 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 27 | 18 | 10 | 8 | 7
Rash (Skin and subcutaneous tissue disorders) | 28 | 24 | 14 | 12 | 7
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 4
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 1
Hypertension (Vascular disorders) | 38 | 10 | 34 | 12 | 13
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 3 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 3 | 0
Anxiety (Psychiatric disorders) | 8 | 6 | 6 | 1 | 6
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 2 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.